CLINICAL TRIAL: NCT07266597
Title: Micropulse Laser Photocoagulation Treatment of Diabetic Macular Edema ; 5 % Versus 15 % Duty Cycle
Brief Title: Micropulse Laser Photocoagulation in Diabetic Macular Edema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Younis Shabaan Aboelhassan, principle investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-7-23MS
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Macular Edema
Keywords: micropulse , diabetic macular edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): will be treated using 5 % duty cycle
  Interventions: Procedure: micropulse laser photocoagulation
- Group B (Active Comparator): will be treated using 15 % duty cycle .
  Interventions: Procedure: micropulse laser photocoagulation

INTERVENTIONS:
Procedure: micropulse laser photocoagulation — micropulse laser photocoagulation in treatment of diabetic macular edema, 5% duty cycle
  Arms: group A
Procedure: micropulse laser photocoagulation — micropulse laser photocoagulation in treatment of diabetic macular edema,15% duty cycle
  Arms: Group B

SUMMARY:
To assess the safety and efficacy of 532 nm subthreshold micropulse laser 5 % duty cycle compared with 15 % duty cycle in treatment of diabetic macular edema .

DETAILED DESCRIPTION:
prospective interventional randomized comparative study that will be conducted on Patients with diabetic retinopathy who Are More than 18 years old with diabetic macular edema with a central retinal thickness < 400 um and best corrected visual acuity between 6/18 and 6/60 .

The participants will be divided randomly into two groups All Patients will receive single session of 532 nm subthreshold micropulse laser ,the following parameters will be used in all cases as follows,spot size : 200-µm ,exposure duration:200-ms ,power : 500-mW

While duty cycle will differ between 2 groups as follows :- Group A : will be treated using 5 % duty cycle . Group B : will be treated using 15 % duty cycle . follow up visits as follows 1 week ,4 weeks 12 weeks after laser therapy .

ELIGIBILITY:
Inclusion Criteria:

Patients with diabetic retinopathy who:

* Are More than 18 years old .
* have diabetic macular edema with a central retinal thickness < 400 um .
* have best corrected visual acuity between 6/18 and 6/60 .

Exclusion Criteria:

* Previous lasered retina , Anti - VEGF injection or vitrectomy .
* Extensive Macular ischemia on FFA .
* Media opacity .
* Associated ocular pathology as glaucoma, CNV (choroidal neovascularization ) , AMD (age related macular degenerations ), epiretinal membrane vitreomacular traction and retinal vein occlusion .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
central macular thickness | 3 months
  assessment of change of central macular thickness before and after laser treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ong J, Selvam A, Maltsev DS. Subthreshold laser systems: a narrative review of the current status and advancements for retinal diseases. Ann Eye Sci. 2022;7:15 .
- [Result] Bodea F, Bungau SG, Bogdan MA, Vesa CM, Radu A, Tarce AG, Purza AL, Tit DM, Bustea C, Radu AF. Micropulse Laser Therapy as an Integral Part of Eye Disease Management. Medicina (Kaunas). 2023 Jul 28;59(8):1388. doi: 10.3390/medicina59081388. PMID 37629677
- [Result] 1. Bakri SJ, Wolfe JD, Regillo CD, Flynn HW, Wykoff CC. Evidence-Based Guidelines for Management of Diabetic Macular Edema. Journal of VitreoRetinal Diseases. 2019;3(3):145-152.